CLINICAL TRIAL: NCT04556929
Title: Improving Fluorescence-guided Brain Tumour Surgery With Ultra-high Sensitivity Imaging
Brief Title: Enhanced Detection in Glioma Excision
Acronym: EDGE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Technical limitations of in-built operative microscope optics
Sponsor: University of Oxford (Other)
Collaborators: Oxford University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 255263
Record Dates: First submitted 2020-07-30; First posted 2020-09-21 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2020-09

CONDITIONS: Glioma
Keywords: 5-Aminolevulinic acid (5-ALA); Malignant glioma; Tumor resection
MeSH Terms: conditions — Glioma | interventions — Biopsy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intraoperative imaging of 5-ALA during tumour resection (Experimental): Participants will undergo 5-ALA guided tumour resection via craniotomy with the aim of achieving maximal safe tumour resection without significant neurological deficit. On completion of tumour resection, digital images will be taken of the resection cavity under blue light using (i) an in-built camera in the operative microscope and (ii) an ultra-high sensitivity camera attached to the side arm of the operative microscope. Biopsies approximately 5x5x5mm in size will then be taken from the anterior, posterior, lateral and inferior areas of the resection cavity which were imaged. These biopsies will be analysed by histopathology to determine the presence of glioma cells.
  Interventions: Diagnostic Test: Intra-operative imaging of 5-ALA fluorescence using ultra-high sensitivity camera; Diagnostic Test: Intra-operative imaging of 5-ALA fluorescence using in-built operative microscope camera; Diagnostic Test: Biopsies

INTERVENTIONS:
Diagnostic Test: Intra-operative imaging of 5-ALA fluorescence using ultra-high sensitivity camera — An ultra-high sensitivity camera attached to the side arm of the operative microscope will be used to take images of the anterior, posterior, lateral and inferior walls of the resection cavity on completion of tumour resection.
Diagnostic Test: Intra-operative imaging of 5-ALA fluorescence using in-built operative microscope camera — In-built camera of the operative microscope will be used to take images of the anterior, posterior, lateral and inferior walls of the resection cavity on completion of tumour resection.
Diagnostic Test: Biopsies — Following image capture, biopsies (approx 5x5x5mm size) will be taken from regions of the anterior, posterior, lateral and inferior walls of the resection cavity corresponding to the imaged areas.

SUMMARY:
The purpose of this study is to determine whether use of an ultra-high sensitivity camera with enhanced imaging technology can be used during surgery to detect areas of brain tissue affected by diffuse glioma, a type of brain cancer.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Male or Female, aged 18 years or above.
* Female patients are not pregnant at time of surgery.
* Patient has consented to craniotomy for suspected glioma of any type with 5-ALA infusion.

Exclusion Criteria:

• Participants are participating in another trial at time of operation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2020-09-21 (Actual); Primary Completion 2021-11-03 (Actual); Study Completion 2021-11-03 (Actual)

PRIMARY OUTCOMES:
Level of tumour fluorescence in images of resection cavity captured during surgery | Intra-operative
  Levels of tumour fluorescence in intra-operative images of the resection cavity taken by the ultra-high sensitivity camera and the in-built camera in the operative microscope will be measured. These fluorescence levels will then be used to calculate the sensitivity and specificity of the in-built camera and ultra-high sensitivity camera to detect glioma tissue.

SECONDARY OUTCOMES:
Duration of operation stages | Intra-operative
  Time points measured will include (i) time from arrival in theatre to start of operation, (ii) total operation duration and (iii) time from acquisition of images to availability of processed images available for the surgeon to view.

CONTACTS AND LOCATIONS:
Overall Officials: Puneet Plaha, MD FRCS, Principal Investigator — University of Oxford
Locations (1):
- John Radcliffe Hospital, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes